CLINICAL TRIAL: NCT07041307
Title: Microvascular Profiling of Nodules in the Thyroid Gland
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Nathalie Sarup Panduro, MD, Rigshospitalet, Denmark
Other Study IDs: SURE-THYROID
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Nodular Disease
Keywords: thyroid nodules; super-resolution ultrasound
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy Participants: Normal Thyroid Gland
- Thyroid Cancer: Malignant Thyroid Nodule
- Hyperfunctioning Nodules: Benign, Hyperfunctioning Thyroid Nodules
- Isofunctioning Nodules: Benign, Isofunctioning Thyroid Nodules
- Hypofunctioning Nodules: Benign, Hypofunctioning Thyroid Nodules

SUMMARY:
The purpose of this study is to examine tiny blood vessels in different thyroid nodules using advanced ultrasound. In the long term, we hope this can help doctors better tell the difference between types of nodules and more accurately decide who may need surgery.

DETAILED DESCRIPTION:
In this study, the investigators use an advanced ultrasound technique called Super-Resolution Ultrasound of Erythrocytes (SURE) to map the microvasculature in the thyroid gland and thyroid nodules. This method provides much higher resolution than conventional ultrasound, allowing us to visualize and measure even the smallest blood vessels.

The investigators aim to explore whether this technique can help differentiate between various types of thyroid nodules - including benign and malignant - and possibly between hyper-, iso-, and hypofunctioning nodules, based on their microvascular characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Written and verbal informed consent to participate in the study
* Patients with hypo-, iso-, or hyperfunctioning thyroid nodules
* Patients referred for thyroid surgery due to suspected malignant nodule (including Bethesda classification groups III, IV, V, and VI)
* Healthy volunteers - generally good health with no chronic illnesses

Exclusion Criteria:

* Pregnancy
* Inability to undergo the examination due to physical or mental limitations
* Desire to opt out of receiving information about new, significant health findings revealed during the study
* Healthy Participants:
* Thyroid disease, including nodules, as well as current or past conditions affecting the thyroid
* Medication that affects thyroid function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited through posters displayed at public institutions such as universities, libraries, and similar locations, as well as via the website https://forskningnu.dk/.
  Patients will be recruited from the Department of Clinical Physiology and Nuclear Medicine, and the Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, both located at Rigshospitalet, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Visualization of the Microvasculature in the Thyroid Gland and Thyroid Nodules | 30 minutes
  With super-resolution ultrasound imaging using the erythrocytes, the investigators will visualize the microvasculature in normal thyroid tissue and different types of thyroid nodules.

SECONDARY OUTCOMES:
Quantification of the Microvasculature | 30 minutes
  Quantification of the thyroid microvasculature and the microvasculature in thyroid nodules. This includes vessel density, vessel diameters, blood flow velocity and vessel distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bachmann Nielsen, Professor PhD dr.med., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Technical University of Denmark, Lyngby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naji MA, Taghavi I, Schou M, Praesius SK, Hansen LN, Panduro NS, Andersen SB, Sogaard SB, Gundlach C, Kjer HM, Tomov BG, Thomsen EV, Nielsen MB, Larsen NB, Dahl AB, Sorensen CM, Jensen JA. Super-Resolution Ultrasound Imaging Using the Erythrocytes-Part II: Velocity Images. IEEE Trans Ultrason Ferroelectr Freq Control. 2024 Aug;71(8):945-959. doi: 10.1109/TUFFC.2024.3411795. Epub 2024 Aug 19. PMID 38857146
- [Background] Arendt Jensen J, Amin Naji M, Kazmarek PraeSius S, Taghavi I, Schou M, Naur Hansen L, Bech Andersen S, Byrholdt Sogaard S, Sarup Panduro N, Mehlin Sorensen C, Bachmann Nielsen M, Gundlach C, Martin Kjer H, Bjorholm Dahl A, Gueorguiev Tomov B, Lind Ommen M, Bent Larsen N, Vilain Thomsen E. Super-Resolution Ultrasound Imaging Using the Erythrocytes-Part I: Density Images. IEEE Trans Ultrason Ferroelectr Freq Control. 2024 Aug;71(8):925-944. doi: 10.1109/TUFFC.2024.3411711. Epub 2024 Aug 19. PMID 38857145
- [Background] Erdogan MF, Anil C, Cesur M, Baskal N, Erdogan G. Color flow Doppler sonography for the etiologic diagnosis of hyperthyroidism. Thyroid. 2007 Mar;17(3):223-8. doi: 10.1089/thy.2006.0104. PMID 17381355
- [Background] Pedersen OM, Aardal NP, Larssen TB, Varhaug JE, Myking O, Vik-Mo H. The value of ultrasonography in predicting autoimmune thyroid disease. Thyroid. 2000 Mar;10(3):251-9. doi: 10.1089/thy.2000.10.251. PMID 10779140
- [Background] Carmeliet P, Jain RK. Angiogenesis in cancer and other diseases. Nature. 2000 Sep 14;407(6801):249-57. doi: 10.1038/35025220. PMID 11001068
- [Background] Arjan JA, Visser M, Zeyl CW, Gerrish PJ, Blanchard JL, Lenski RE. Diminishing returns from mutation supply rate in asexual populations. Science. 1999 Jan 15;283(5400):404-6. doi: 10.1126/science.283.5400.404. PMID 9888858
- [Background] Russ G, Bonnema SJ, Erdogan MF, Durante C, Ngu R, Leenhardt L. European Thyroid Association Guidelines for Ultrasound Malignancy Risk Stratification of Thyroid Nodules in Adults: The EU-TIRADS. Eur Thyroid J. 2017 Sep;6(5):225-237. doi: 10.1159/000478927. Epub 2017 Aug 8. PMID 29167761
- [Background] Knudsen N, Bulow I, Jorgensen T, Laurberg P, Ovesen L, Perrild H. Goitre prevalence and thyroid abnormalities at ultrasonography: a comparative epidemiological study in two regions with slightly different iodine status. Clin Endocrinol (Oxf). 2000 Oct;53(4):479-85. doi: 10.1046/j.1365-2265.2000.01121.x. PMID 11012573
- See also: Related Info — https://www.cancer.dk/skjoldbruskkirtelkraeft-thyreoideacancer/fakta/statistik/
- See also: Related Info — https://endocrinology.dk/nbv/thyroideasygdomme/udredning-af-knuden-i-glandula-thyreoidea/